CLINICAL TRIAL: NCT05098509
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled Study of RAD011 (Cannabidiol Oral Solution) for the Treatment of Patients With Prader- Willi Syndrome
Brief Title: A Study to Assess RAD011 (Cannabidiol Oral Solution) for the Treatment of Participants With Prader-Willi Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to a change in corporate priorities, this study was voluntarily terminated by the Sponsor for reasons other than safety
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCOUT-015
Record Dates: First submitted 2021-09-22; First posted 2021-10-28 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RAD011 40 milligrams per kilogram (mg/kg) (Active Comparator): Participants were administered 40 mg/kg of RAD011 orally daily with food.
  Interventions: Drug: RAD011
- RAD011 20 mg/kg (Active Comparator): Participants were administered 20 mg/kg of RAD011 orally daily with food.
  Interventions: Drug: RAD011
- RAD011 10 mg/kg (Active Comparator): Participants were administered 10 mg/kg of RAD011 orally daily with food.
  Interventions: Drug: RAD011
- Placebo (Placebo Comparator): Participants were administered a placebo matching to RAD011, orally daily with food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD011 — Cannabidiol Oral Solution (containing synthetic cannabidiol)
  Arms: RAD011 10 mg/kg; RAD011 20 mg/kg; RAD011 40 milligrams per kilogram (mg/kg)
Drug: Placebo — Matching Placebo for RAD011
  Arms: Placebo

SUMMARY:
This was a study investigating RAD011 in participants diagnosed with Prader-Willi Syndrome (PWS). The primary objective of the Phase 2 part of this study was to assess the safety and tolerability of multiple dose levels of RAD011 in order to select 1 or 2 dose level(s) for further evaluation in the Phase 3 part of the study. In Phase 3, the primary objective was to assess the effect of RAD011 on hyperphagia-related behavior in participants with PWS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 8 and 65 years of age (inclusive) at Screening.
* Genetically confirmed diagnosis of PWS. Documentation of genetically confirmed diagnosis of PWS is acceptable.
* The same caregiver is available to complete the questionnaire throughout the duration of the study.
* After completion of the Tolerability period, participants will have a mean Hyperphagia Questionnaire for Clinical Trials (HQ-CT) score ≥13 and a decrease of HQ-CT score no more than 7 during Tolerability (run-in) period.
* If receiving growth hormone, psychotropic therapy, metabolic treatments that could affect appetite (including metformin), and other treatment including thyroid hormone, must be on the same medication and dose for at least 90 days prior to consent/assent

Exclusion Criteria:

* Known use of cannabis or cannabinoid containing products (including topical products) within 90 days prior to consent/ assent.
* Use of prescription or over-the-counter weight loss agents within 90 days prior to consent/assent.
* Implementation of new food or environmental restrictions within 90 days of consent/ assent.
* If living in a group home, participant spends less than 25 waking hours with their caregiver per week.
* Uncontrolled chronic conditions (diabetes, sleep apnea, etc.) as determined by the Investigator.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - Maimonides Medical Center, Brooklyn, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - MultiCare Institute for Research & Innovation, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 4 participants were randomized and received at least 1 dose of study drug. No participants were randomized to the placebo group. The 4 participants were randomized in Phase 2 of the study and due to premature termination of the study, phase 3 was not conducted. None of the enrolled participants completed the study due to the study being terminated prematurely.
Groups:
- RAD011 10 Milligrams Per Kilogram (mg/kg): Participants were administered 10 mg/kg of RAD011 orally daily with food.
- RAD011 40 mg/kg: Participants were administered 40 mg/kg of RAD011 orally daily with food.
Period: Overall Study
Arm/Group | RAD011 10 Milligrams Per Kilogram (mg/kg) | RAD011 20 mg/kg | RAD011 40 mg/kg | Placebo
Started | 1 | 1 | 2 | 0
Received 1 Dose of Study Drug | 1 | 1 | 2 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Early study termination | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Population included all randomized participants who received at least 1 dose of study drug. Due to the small sample size, data was not reported for confidentiality reasons.
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | NA [NA to NA] — Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons. | NA [NA to NA] — Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons. | NA [NA to NA] — Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons. | NA [NA to NA] — Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size for this baseline characteristic, data was not reported for confidentiality reasons.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 34 in the Hyperphagia Questionnaire for Clinical Trials (HQ-CT) Questionnaire
Description: The HQ-CT measures hyperphagia by Prader-Willi syndrome (PWS)-specialized clinicians. The HQ-CT generates a score ranging from 0 to 36, where a higher score represents more severe abnormal food related behaviors.
  The change from baseline was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: Baseline, Week 34
Population: Due to the premature termination of the study, no efficacy analyses were conducted. Therefore, no data was collected for this outcome measure.
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline to Week 34 in Prader-Willi Syndrome (PWS)- Associated Irritability Using the Aberrant Behavior Checklist (ABC) Questionnaire - Irritability Subscale (ABC-I)
Description: The ABC questionnaire is an informant-rated questionnaire assessing severity of behavioral symptoms. The Irritability subscale of the ABC covers symptoms such as agitation, aggression, meltdowns, and self-harm. The ABC-I contains 15 items and each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). The total score is the sum of individual items scores which ranges from 0 (no problem) to 45 (severe problem), with higher score indicating more severe condition.
Time Frame: Baseline, Week 34
Population: as for outcome 1
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline to Week 34 in Hyperphagia as Measured by the Clinician Global Impression of Change (CGI-C)
Description: The CGI-C of hyperphagia is a single-item, clinician-rated measure, assessing the clinician's impression about changes in the patient's hyperphagia condition since the start of taking the study medication at the initiation of the Tolerability Period. The CGI-C of hyperphagia utilizes a 5-point response scale: 1=Much better; 2=A little better; 3=No change; 4=A little worse; 5=Much worse. Higher scores mean a worse outcome.
Time Frame: Baseline, Week 34
Population: as for outcome 1
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline to Week 34 in Hyperphagia as Measured by the Clinician Global Impression of Severity (CGI-S)
Description: The CGI-S of hyperphagia is a single-item, clinician-rated measure, assessing the clinician's impression of the severity of a patient's hyperphagia condition. The CGI-S of hyperphagia utilizes a 5-point response scale: 1=None; 2=Mild; 3=Moderate; 4=Severe; 5=Very Severe. Higher scores mean a worse outcome.
Time Frame: Baseline, Week 34
Population: as for outcome 1
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to 68 days (maximum duration from treatment to early termination)
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | RAD011 10 mg/kg | RAD011 20 mg/kg | RAD011 40 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD011 10 mg/kg (N=1) | RAD011 20 mg/kg (N=1) | RAD011 40 mg/kg (N=2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study has been voluntarily terminated by the sponsor due to change in corporate priorities, for reasons other than safety. Due to early termination of study, no efficacy analyses were done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05098509/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05098509/SAP_001.pdf